CLINICAL TRIAL: NCT02902120
Title: Host Mechanisms Involved in Achieving SVR Using Grazoprevir and Elbasvir in Treatment of Chronic Hepatitis C in Patients With CKD Before and After Renal Transplantation
Brief Title: HCV Treatment Immune Response With Grazoprevir/Elbasvir Before or After Renal Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jennifer Husson, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00071069
Record Dates: First submitted 2016-08-19; First posted 2016-09-15 (Estimated); Results first posted 2022-11-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis C; Renal Insufficiency, Chronic; Disorder of Transplanted Kidney
MeSH Terms: conditions — Hepatitis C; Renal Insufficiency, Chronic | interventions — elbasvir; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Post-transplant (Experimental): This arm will evaluate the treatment of patients with HCV and chronic kidney disease (GFR <50) who have had a kidney transplant using grazoprevir and elbasvir.
  Interventions: Drug: Post-transplant Grazoprevir and Elbasvir

INTERVENTIONS:
Drug: Post-transplant Grazoprevir and Elbasvir — Treatment will be started in the post-transplant patients on day 0 with the combination pill zepatier, containing grazoprevir 100mg/elbasvir 50mg by mouth once daily. The medications will be continued for a total of 12 weeks (16 weeks if resistance mutations, RAVs, are detected)
  Other Names: Zepatier

SUMMARY:
The purpose of this study is to determine whether patients treated for chronic hepatitis C (HCV) with zepatier (grazoprevir/elbasvir) prior to kidney transplant will have a stronger immune response compared to patients treated after kidney transplant. 25 patients with chronic kidney disease (CKD) and HCV will be treated with zepatier and 25 kidney transplant recipients with chronic kidney disease will be treated with zepatier. Blood markers of immune function will be monitored in both groups to determine their response to therapy.

DETAILED DESCRIPTION:
The study will be a pilot, prospective, single-center, open-label, non-randomized, non-controlled, parallel clinical trial. 25 HCV genotype 1 infected patients post transplant will be enrolled in the study. Recruitment will be conducted through the renal transplant and nephrology outpatient clinics at the University of Maryland.

The post-transplant cohort will include renal transplant recipients of both living donor and deceased donor organs infected with HCV prior to their transplantation with GFRs <50 with active HCV viremia. These patients will be recruited from the University of Maryland's multidisciplinary transplant nephrology clinic or infectious disease clinic.

Screening All patients will be screened at the Institute of Human Virology (IHV) Clinical Research Unit. At this visit, all patients will have screening labs drawn and a history and physical examination performed. Additional requirements will be genotype testing prior to enrollment, but after transplant and disease staging within 12 months of enrollment by liver biopsy, elastography, or biochemical testing. For those who do not have a genotype or disease staging within the specified time frame, genotyping and elastography will be repeated as part of the study screening work up. Eligibility will be determined based upon these results within 6 weeks of starting the study drugs.

Given the reduced efficacy of this regimen in patients with genotype 1a with the presence of baseline NS5A resistance-associated variants (RAVs), the investigators will screen patients for RAVs in patients with HCV genotype 1a at the time of enrollment. Any patient with genotype 1a HCV found to have NS5A RAVs will undergo 16 weeks of therapy according to current treatment guidelines.

Starting therapy Study drugs will be administered starting on day 0 after a history and physical examination is performed and safety labs are checked. All patients will sign an informed consent as approved by our Institutional Review Board (IRB) prior to administration of study drugs.

Study visits during treatment Patients will be followed every 4 weeks while they are receiving study drugs. HCV viral load (VL), safety labs and hepatic panel will be performed at each of these visits. Patients will also be advised about study adherence and monitored for adverse events.

Safety and adverse event monitoring At each study visit, research nurses will inquire about adverse events that may or may not be related to study drugs. Any unfavorable medical occurrences will be recorded, whether or not considered related to the patient's participation in the research, temporally associated with the patient's participation in the research. Adverse events (AEs) classified as grade 3 or higher will be reported to the IRB and principal investigator. Any grade 3 or 4 AEs and all serious adverse events (SAEs) will be reviewed as they occur by the study team.

Safety labs will also be drawn at these visits. Levels of immunosuppressive agents will also be determined at these visits as appropriate. The need for dose modification of the patient's immunosuppression in the time between visits will be recorded.

End of treatment visit Patients will be seen 12 weeks after starting study drugs (or 16 weeks in the case of genotype 1a patients with baseline NS5A RAVs) for an end of study visit. HCV VL, safety labs and hepatic panel will be performed at this visit. Patients will also be counseled about study adherence and the investigators will inquire about adverse events.

Post treatment follow up visits Patients will be followed every 4 weeks for 12 weeks after they complete treatment. HCV VL, safety labs and a hepatic panel will be performed at these visits.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of screening
* Have stable renal function for one month (30 days) prior to enrollment
* Have Chronic HCV infection prior to transplantation with documented HCV viremia ≥ 1,000 IU/ml at screening and either documented HCV Ab positivity or HCV viremia ≥ 1,000 IU/ml at least 6 months prior to enrollment.
* Documented genotype 1 HCV infection prior to enrollment and after their transplant in the post-transplantation cohort
* HCV disease staging within 12 months prior to enrollment by liver biopsy, transient elastography, or biochemical testing
* Be able to give informed consent and comply with study guidelines
* Women of childbearing age will be required to have a negative pregnancy test at enrollment and use birth control throughout the duration of treatment.

Inclusion Criteria Specific to the Pre-transplant Arm

Patients will either be:

* On the transplant waiting list followed by the University of Maryland's nephrology clinic or the Baltimore VA's nephrology clinic
* On chronic hemodialysis not yet on the transplant list and followed in the University's hemodialysis center or in the University's nephrology clinic
* Have chronic kidney disease with GFR <50

Inclusion Criteria Specific to the Post-transplant Arm

• Patients will have undergone renal transplantation no greater than five years prior to enrollment and will be followed in our University's nephrology and infectious disease clinic. They will all have stable renal function at the time of enrollment.

Exclusion Criteria:

* Documented positive hepatitis B (HBV) surface antigen, and/or HBV DNA prior to enrollment
* Any prior exposure to HCV protease inhibitor therapy
* HIV co-infection if on a protease inhibitor based regimen
* Increase in creatinine of 15% or greater within one month (30 days) of the screening visit
* Evidence of hepatocellular carcinoma at the time of enrollment
* Liver disease caused by an etiology other than HCV
* F4 or decompensated cirrhotic patients
* Child Pugh class B or C
* AST or ALT >350 within 6 months prior to enrollment
* Albumin < 3g/dL at the time of enrollment
* Platelet count < 75 at the time of enrollment
* History of clinically significant allergy or adverse event with protease inhibitors
* Evidence of the acquisition of HCV at the time of or after transplantation
* Pregnant or breastfeeding women
* Cyclosporine; St. John's Wort; Efavirenz; Phenytoin; Carbamazepine; Bosentan; HIV protease inhibitors; modafinil; ketoconazole; or rifampin use within 7 days of enrollment
* Coadministration of more than 20 mg atorvastatin; 10 mg rosuvastatin; 20 mg of fluvastatin, lovastatin or simvastatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Husson, MD, Principal Investigator — University of Maryland School of Medicine, Institute of Human Virology
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification will be shared.
Supporting Information: Study Protocol
Time Frame: Data will be available immediately upon publication for a duration of 5 years following publication.
Access Criteria: Investigators who provide a methodologically sound proposal to achieve the aims in the approved proposal.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post-transplant
Started | 21
Completed | 20
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Post-transplant
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.65 (8.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Fibrosis Stage [Count of Participants; unit: Participants] — Fibrosis staging was done within 12 months prior to enrollment by liver biopsy, transient elastography using Fibroscan or biochemical testing using FibroTest. These tests produced results corresponding to a fibrosis stage with a fibrosis stage 0-1 being less severe and 2-3 being more severe fibrosis. Fibrosis stage 4, being the most severe/cirrhosis, was excluded from the study.
  Six participants had disease staging done by liver biopsy, 6 participants by transient elastography using Fibroscan, and 9 participants by biochemical testing by FibroTest.
  Participants
    Fibrosis Stage 0-1 | 12
    Fibrosis Stage 2-3 | 9
HCV-positive donor [Count of Participants; unit: Participants] | 19
HCV genotype post-transplant [Count of Participants; unit: Participants] — HCV genotype as measured by a serum HCV genotype test, prior to HCV treatment. Genotype 1 was required for inclusion based upon the treatment recommendations for elbasvir/grazoprevir in genotype 1 at the time. Data was further used to detect genotype 1a which required additional testing to ensure no NS5a resistance associated variants (RAVs) were present which may impact the duration of treatment.
  Participants
    Genotype 1a | 14
    Genotype 1b | 7
Median baseline HCV RNA level [Median (Full Range); unit: Log international units/mL] | 6.24 [5.56 to 6.65]
Time from transplant [Mean (Full Range); unit: days] | 117 [44 to 321]

OUTCOME MEASURES:

1. Primary Outcome: SVR 12
Description: Sustained virologic response (SVR) will be assessed by measuring the quantitative HCV viral load 12 weeks after completing treatment. This will be a measure of circulating HCV virus in participants off therapy, 12 weeks after finishing treatment, to determine the durability of the response to the treatment.
Time Frame: This will be measured at post-treatment week 12 (study week 24 or week 28 for those with resistance mutations)
Measure: Count of Participants; unit: Participants
Arm/Group | Post-transplant
Number analyzed (Participants) | 21
Participants
  Number achieved SVR12 | 19
  Number failed treatment | 1
  Number missing SVR12 data | 1

2. Secondary Outcome: Change in T Cell Response
Description: The study will involve measuring the change in T cell response by analyzing the frequency of exhaustion markers PD-1 and activation markers ICOS, CD38, CD69 at day 0, week 4, and week 12.
Time Frame: This will be collected at day 0, week 4, and week 12
Population: This study was amended to eliminate the comparator arm and focus on clinical outcomes including SVR12. No subjects were recruited in this arm, so no data was collected or is available.
Measure: Mean (Standard Deviation); unit: percentage of expressing cells
Arm/Group | Post-transplant
Number analyzed (Participants) | 6
percentage of expressing cells
  PD-1 day 0 | 29.15 (15.21)
  PD-1 week 4 | 21.83 (14.52)
  PD-1 week 12 | 20.5 (8.91)
  ICOS day 0 | 12.73 (7.92)
  ICOS week 4 | 6.14 (5.65)
  ICOS week 12 | 5.03 (2.81)
  CD38 day 0 | 10.86 (4.81)
  CD38 week 4 | 5.97 (4.43)
  CD38 week 12 | 6.73 (4.48)
  CD69 day 0 | 0.98 (0.60)
  CD69 week 4 | 0.43 (0.26)
  CD69 week 12 | 0.75 (0.54)

3. Secondary Outcome: Change in T Cell Immunophenotypes
Description: The study will involve measuring the change in T cell immunophenotypes
Time Frame: This will be collected at day 0, week 4, and week 12
Population: This study was amended to eliminate the comparator arm and focus on clinical outcomes including SVR12. No subjects were recruited in this arm, so no data was collected or is available.
  The frequency of CD4+ and CD8+ effector memory, naïve, central memory and terminally differentiated effector memory cell populations were compared from day 0 to week 4 on treatment.
Measure: Mean (Standard Deviation); unit: percentage of expressing cells
Arm/Group | Post-transplant
Number analyzed (Participants) | 9
percentage of expressing cells
  CD4+CCR7-CD45RO+ EM day 0 | 70.64 (17.48)
  CD4+CCR7-CD45RO+ EM week 4 | 65.4 (11.17)
  CD4+CCR7-CD45RO+ EM week 12 | 65.1 (13.29)

4. Secondary Outcome: Quantification of Antiviral Cytokines
Description: The study will involve measuring interferon gamma and TNF alpha levels
Time Frame: This will be collected at day 0 and week 4
Population: This study was amended to eliminate the comparator arm and focus on clinical outcomes including SVR12. No subjects were recruited in this arm, so no data was collected or is available.
  Analysis was done comparing IFN gamma and TNF alpha from day 0 to week 4.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Post-transplant
Number analyzed (Participants) | 19
pg/mL
  IFN gamma day 0 | 9.67 (7.12)
  IFN gamma week 4 | 7.26 (6.19)
  TNF alpha day 0 | 7.26 (2.74)
  TNF alpha week 4 | 4.45 (3.55)

5. Secondary Outcome: Safety as Assessed by Adverse Event Monitoring, Including Routine Lab Work
Description: Safety will be assessed by adverse event monitoring, including routine lab work
Time Frame: This will be measured at day 0, weeks 2, 4, 8, 12 (and 16 if resistance mutations are present)
Measure: Count of Participants; unit: Participants
Arm/Group | Post-transplant
Number analyzed (Participants) | 21
Participants
  Any Adverse Event: Yes | 21
  Any Adverse Event: No | 0
  Any Serious Adverse Event: Yes | 6
  Any Serious Adverse Event: No | 15
  Decrease in eGFR >30% from baseline: Yes | 4
  Decrease in eGFR >30% from baseline: No | 17
  Elevated tacrolimus level while on treatment: Yes | 13
  Elevated tacrolimus level while on treatment: No | 8

6. Secondary Outcome: Kidney Function
Description: Clinical review using labs and the patient's chart will be performed for change in kidney graft function by change in eGFR or creatinine
Time Frame: This will be measured at day 0, treatment week 2, treatment week 4, treatment week 8, treatment week 12, ( treatment week 16, if applicable), post-treatment week 4 (week 16/20), and post-treatment week 12 (week 24/28)
Measure: Count of Participants; unit: Participants
Arm/Group | Post-transplant
Number analyzed (Participants) | 21
Participants
  Increase in Cr >30% on treatment: yes | 5
  Increase in Cr >30% on treatment: no | 16
  Decrease eGFR >30%: yes | 4
  Decrease eGFR >30%: no | 17

7. Secondary Outcome: Kidney Allograft Rejection
Description: Clinical review using labs and the patient's chart will be performed for documented episodes of kidney rejection
Time Frame: This will be measured at post-treatment week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Post-transplant
Number analyzed (Participants) | 21
Participants
  Borderline acute cellular rejection | 1
  Mild antibody mediated rejection | 1
  No rejection | 19

ADVERSE EVENTS:
Time Frame: Adverse event information was collected throughout the subjects participation in the study, from screening through post-treatment week 12 at the following timepoints: day 0, treatment week 2, treatment week 4, treatment week 8, treatment week 12, ( treatment week 16, if applicable), post-treatment week 4 (week 16/20), and post-treatment week 12 (week 24/28).
Arm/Group | Post-transplant
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-transplant (N=21)
Nausea, vomiting (Gastrointestinal disorders) | 3 (3) — Nausea, vomiting resulting in hospitalization
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Shortness of breath resulting in hospitalization
CMV Viremia (Infections and infestations) | 1 (1) — CMV Viremia resulting in hospitalization
Decreased appetite (Gastrointestinal disorders) | 2 (2) — Decreased appetite and intake leading to hospitalization
UTI, sepsis (Infections and infestations) | 1 (1) — UTI, sepsis with hospitalization
Diarrhea (Gastrointestinal disorders) | 1 (1) — Diarrhea resulting in hospitalization
acute kidney injury (Renal and urinary disorders) | 1 (1) — acute kidney injury resulting in hospitalization
Fatigue (General disorders) | 1 (1) — Fatigue with nausea, vomiting, diarrhea and acute kidney injury leading to hospitalization
Diabetic ketoacidosis (Endocrine disorders) | 1 (1) — DKA with shingles requiring hospitalization
Shingles (Infections and infestations) | 1 (1) — DKA with shingles requiring hospitalization
URI (Infections and infestations) | 1 (1) — URI requiring hospitalization
Community acquired pneumonia (Infections and infestations) | 1 (1) — CAP requiring hospitalization
Acute kidney injury (Renal and urinary disorders) | 1 (1) — AKI requiring hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-transplant (N=21)
Fatigue (General disorders) | 9 (9)
Elevated tacrolimus level (Renal and urinary disorders) | 17 (73)
Elevated creatinine or AKI (Renal and urinary disorders) | 6 (21) — elevated Cr >30% baseline or a diagnosis of AKI
Low platelets (Blood and lymphatic system disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5) — Diarrhea not requiring hospitalization
nausea, vomiting (Gastrointestinal disorders) | 1 (1) — nausea, vomiting not requiring hospitalization
UTI (Infections and infestations) | 4 (5)
candida infection (Infections and infestations) | 3 (5) — oral thrush, esophagitis
CMV viremia, syndrome (Infections and infestations) | 4 (4)
anemia (Blood and lymphatic system disorders) | 1 (1)
shingles (Infections and infestations) | 2
Tremor (Nervous system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) — Low WBC count
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Decreased Tacrolimus levels (Investigations) | 19 (138)
Microalbuminuria (Renal and urinary disorders) | 3 (3)
ankle swelling (Vascular disorders) | 1 (1)
Elevated WBCs (Blood and lymphatic system disorders) | 1 (1)
seasonal allergies (Immune system disorders) | 1 (1)
pruritis (Immune system disorders) | 1 (1)
dry cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
decreased appetite (General disorders) | 1 (1)
orchitis (Reproductive system and breast disorders) | 1 (1)
mild antibody mediated rejection (Immune system disorders) | 1 (1)
increased glucose (Endocrine disorders) | 1 (2)
Groin strain or pain (Musculoskeletal and connective tissue disorders) | 2 (2)
fall (Nervous system disorders) | 2 (2)
Elevated Blood Pressure (Cardiac disorders) | 1 (3)
Hypotension (Cardiac disorders) | 1 (1)
osteoporosis (Endocrine disorders) | 1 (1)
pyuria (Renal and urinary disorders) | 1 (1)
cold sweats (Endocrine disorders) | 1 (1)
neuropathy (Nervous system disorders) | 2 (2)
Stye (Infections and infestations) | 1 (1)
URI, pharyngitis, rhinitis, bronchitis (Infections and infestations) | 4 (6)
indigestion, GERD (Gastrointestinal disorders) | 1 (1)
muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
otitis media (Ear and labyrinth disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT02902120/Prot_SAP_000.pdf